CLINICAL TRIAL: NCT06503159
Title: Hippocampal Network Changes Following Mindfulness Training in Tobacco Vaping Adolescents
Brief Title: Hippocampal Network Changes Following Mindfulness Training in Tobacco Vaping Adolescents in an Open-label, Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left NIH.
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 10001855; 001855-DA
Record Dates: First submitted 2024-07-13; First posted 2024-07-16 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Vaping Teens; Healthy Volunteers
Keywords: Natural History; Teen; Nicotine; Vape
MeSH Terms: conditions — Vaping | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-based Stress Reduction (MBSR) Program (Experimental): This protocol will use fMRI and in-person and technology-delivered mindfulness-based stress reduction (MBSR) training to elucidate neurobehavioral correlates of regular nicotine vaping in adolescents compared to non-vaping adolescents, and changes in these correlates after MBSR training.
  Interventions: Behavioral: Mindfulness-based Stress Reduction (MBSR) Program

INTERVENTIONS:
Behavioral: Mindfulness-based Stress Reduction (MBSR) Program — The study intervention is a 9-week MBSR intervention once per week in-person or remotely (via an NIH approved remote platform used in compliance with policy, including HRPP Policy 303). The MBSR will be delivered to groups of 8-12 participants. Only the vaping adolescents will receive MBSR training.

SUMMARY:
The purpose of this translational bench-to-bedside study is to examine the neurobiological effects of an evidence-based technology-delivered mindfulness training (MT) program on vaping-related rsFC alterations in hippocampal networks and testing whether changes in rsFC ((Delta)rsFC) in these networks predict reduction in tobacco vaping behaviors in adolescents. The study also aims to test the accessibility and feasibility of using this mindfulness-based stress reduction (MBSR) platform as an implementation for widespread MT in adolescents....

DETAILED DESCRIPTION:
Study Description:

This protocol will use fMRI and in-person and technology-delivered mindfulness-based stress reduction (MBSR) training to elucidate neurobehavioral correlates of regular nicotine vaping in adolescents compared to non-vaping adolescents, and changes in these correlates after MBSR training. Our central hypothesis is that nicotine vaping in adolescents will be associated with impaired hippocampal connectivity with large-scale brain networks (e.g., Executive Control network (ECN), Default Mode Network (DMN), Salience Network (SN)) involved in cognitive control and emotion regulation and decreased state transitions (measured via dynamic resting state functional connectivity (rsFC)); and that MBSR training will increase hippocampal connectivity to ECN and alter time in state and state transitions in frequent vaping adolescents, with these rsFC changes predicting changes in vaping behavior.

Objectives:

Primary Objectives:

1. To characterize static and dynamic rsFC of hippocampal networks in frequent nicotine vaping adolescents compared to non-vaping adolescents.
2. To characterize rsFC changes in hippocampal networks following an in-person and technology-delivered MBSR training program in frequent nicotine vaping adolescents.

Secondary Objectives:

* To assess engagement with a smoking cessation app and changes in vaping behavior, emotion and cognition in the 3 months following MBSR training.
* To assess differences between vaping and non-vaping teens pre- and post-MBSR training on other measures of network connectivity.

Endpoints:

Primary Endpoints:

* (1) Seed-based rsFC between hippocampal seed regions and large-scale brain networks (DMN, ECN, SN) and dynamicrsFC measures in 40 nicotine vaping and 40 non-vaping youth.
* (2) Seed-based rsFC between hippocampal seed regions and large-scale brain networks (DMN, ECN, SN) and dynamicrsFC measures within the nicotine vaping group Pre/Post MBSR training.

Secondary Endpoint:

* Engagement with MBSR training and post-training Cravingto- Quit app and change scores for other behavioral measure (e.g. vaping, emotion regulation).
* rsFC from seeds such as dorsal anterior cingulate.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

Non-Vaping group:

1. For adolescents aged 17 and under, parental/guardian informed consent to participate in the study
2. English language fluency
3. Males and females; Age 13-18 enrolled in grades 9-12, or the summer after graduation.
4. No MRI contraindications
5. No evidence of current psychosis, mania, or significant suicidality
6. If on medication for depression, anxiety or ADHD, dose has been stable for 3 months
7. No DSM-5 diagnosis of moderate or severe SUD related to a psychoactive substance, including tobacco, in the past year
8. Access to necessary resources for participating in a technology-based intervention, which includes smartphone ownership for this study
9. No use of nicotine more than 5 times in their life, and none at all in the last 30 days prior to enrollment.

Vaping group:

1. For adolescents aged 17 and under, parental/guardian informed consent to participate in the study
2. English language fluency
3. Males and females; Age 13-18 enrolled in grades 9-12, or the summer after graduation.
4. No MRI contraindications
5. No evidence of current psychosis, mania, or significant suicidality
6. If on medication for depression, anxiety or ADHD, dose has been stable for 3 months
7. No DSM-5 diagnosis of moderate or severe SUD related to another psychoactive substance (other than tobacco) in the past year
8. Vape a nicotine containing product at least 10 days in the past 30 days
9. Access to necessary resources for participating in a technology-based intervention, which includes smartphone ownership for this study

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study based on self and or parent-report unless otherwise noted:

Vaping or Non-Vaping Group:

1. Chronic medical conditions associated with cerebral blood flow abnormalities per PI/MAI determination after review of the medical history.
2. Neurological conditions that may interfere with MRI data quality per PI/MAI determination after review of the medical history.
3. Neurodevelopmental disorders that are likely to significantly affect data in the judgment of the MAI/PI
4. Non-penetrating traumatic brain injury with loss of consciousness > 30 minutes or significant sequalae persisting longer than 2 weeks or any penetrating traumatic brain injury.
5. Changing dose of psychotropic medication in past 3 months
6. Current regular meditation or yoga practice averaging >10 min/day for >2 days per week
7. Pregnancy, self-report upon protocol entry, but by urine test prior to MRI scan.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2025-05-07 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
To characterize rsFC changes ((Delta)rsFC) in hippocampal networks and d-rsFC following a technology-delivered MBSR program in nicotine vaping adolescents. | 5.5-7 months
  Hippocampal connectivity and d-rsFC measures are related to both nicotine exposure and MBSR training
To characterize static and dynamic rsFC differences in hippocampal networks related to nicotine vaping in adolescents. | 5.5-7 months
  Hippocampal networks are related to nicotine exposure, especially in adolescence.

SECONDARY OUTCOMES:
To assess other imaging metrics such as resting connectivity from alternative sites related to mindfulness meditation and nicotine dependence (e.g., dACC) between vaping and non-vaping teens and pre-/post-MBSR tr | 5.5-7 months
  These metrics will provide a fuller understanding of teen vaping and the effects of MBSR training.
To assess engagement with a smoking cessation app and changes in various behaviors following MBSR training. | 5.5-7 months
  Understanding feasibility and acceptability as well as efficacy is important in assessing potential for development of MBSR training as a new therapeutic intervention for vaping-related TUD in youth.

CONTACTS AND LOCATIONS:
Overall Officials: Betty Jo Salmeron, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No